CLINICAL TRIAL: NCT02687516
Title: Treatment of Severely Obese Children and Adolescents in Common Health Care Settings: An Effectiveness Study Employing "Family-based Behavioral Social Facilitation Treatment"
Brief Title: Treatment of Severely Obese Children and Adolescents Employing "Family-based Behavioral Social Facilitation Treatment"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Petur B Juliusson, MD/PhD, University of Bergen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1300/REK Vest
Record Dates: First submitted 2014-02-21; First posted 2016-02-22 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Childhood Obesity
Keywords: Treatment; Child; Obesity; Behavioral treatment
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-based behavioral social facilitation therapy. (Experimental): The FBSFT condition includes 17 weekly family-based treatment sessions at the hospital obesity clinic followed by monthly follow-up sessions with their local nurse and follow-up sessions at the hospital every third month for 2 years.The treatment targets both child and parent life-style; eating habits, physical activity, sedentary activity and sleep habits. Behavior modification techniques are systematically employed; such as self-monitoring, goal setting, reward systems, problem solving and stimulus control. In addition, FBSFT focuses on facilitating lifestyle change across different settings (family, friends, school and community) and harnessing social support for healthy habits, which is considered important for long-term weight control.
  Interventions: Behavioral: Family-based behavioral social facilitation therapy
- Treatment as usual (Active Comparator): The TAU condition involves an assessment day with the multidisciplinary team (pediatrician, dietician, physical therapist and psychologist) at the hospital obesity clinic. Further a session with the nurse at the hospital clinic making a plan for behavioral lifestyle changes followed by monthly follow-up sessions with their local nurse and follow-up sessions at the hospital clinic every third month for 12 months. After 12 months they will be offered treatment by family-based behavioral social facilitation therapy (as in the other treatment arm).
  Interventions: Behavioral: TAU - Treatment as usual

INTERVENTIONS:
Behavioral: Family-based behavioral social facilitation therapy — Family-based Behavioral Social Facilitation Treatment (FBSFT) is founded on the principles of standard family-based behavioural therapy for obesity. FBSFT targets life-style behaviors (diet, physical activity and sedentary activity) in a family setting. FBSFT includes some cognitive elements that are considered important in relation to behavioural change for instance problem solving and cognitive restructuring. FBSFT has an intensive treatment phase including weekly family meetings with therapists over 17 consecutive weeks. Further monthly or bi-weekly follow-up sessions with a focus on social facilitation and maintenance of healthy habits are recommended. The dietary guidance of FBSFT is based on the "Traffic light diet" in which foods are organized into GREEN, YELLOW and RED groups. Activity guidance of FBSFT uses the same system: GREEN activities have the highest intensity and should be engaged in most often, YELLOW activities sometimes, and RED activities.
  Arms: Family-based behavioral social facilitation therapy.
Behavioral: TAU - Treatment as usual — This is the default treatment at the obesity clinic. After initial evaluation by paediatrician, nurse, nutritionist and physiotherapist, a "contract" is written including weight goal, nutritional plan and activity plan. Follow up monthly in primary Health care and every 3rd month at the obesity clinic.
  Arms: Treatment as usual

SUMMARY:
This study aims to evaluate the effectiveness of Family-based behavioral social facilitation therapy (FBSFT) in the treatment of severe obesity in children and adolescents compared to treatment as usual (TAU). The FBSFT condition includes 17 weekly family-based treatment sessions at the hospital obesity clinic followed by monthly follow-up sessions with their local nurse and follow-up sessions at the hospital every third month for 2 years. The treatment targets both child and parent life-style; eating habits, physical activity, sedentary activity and sleep habits. Behavior modification techniques are employed; such as self-monitoring, goal setting, reward systems, problem solving and stimulus control. In addition, FBSFT focuses on facilitating lifestyle change across different settings (family, friends, school and community) and harnessing social support for healthy habits, which is considered important for long-term weight control. The TAU condition involves an assessment day with the multidisciplinary team (pediatrician, dietician, physical therapist and psychologist) at the hospital obesity clinic. Further a session with the nurse at the hospital clinic making a plan for behavioral lifestyle changes followed by monthly follow-up sessions with their local nurse and follow-up sessions at the hospital clinic every third month for one year.

SAMPLE AND STUDY DESIGN. The sample will consist of children and adolescents (aged 6-18) referred to the Obesity Outpatient Clinic at Haukeland University Hospital. Criteria for admission to the clinic is an (IOTF) isoBMI of > 35, or a isoBMI > 30 with obesity related co-morbidity. Based on current clinic data, estimations suggest that about 60 families of children with severe obesity will be referred to the Obesity Outpatient Clinic every year and be offered treatment. Recruitment will start in February 2014 and will continue in 2015 and 2016. After consenting to participation and completion of the initial assessments the families will be randomized to either FBSFT or treatment as usual (TAU). After one year the families randomized to TAU will be offered the FBSFT treatment. Measurement points for the most important outcome measures will be pre-treatment, post-treatment (at approximately 6 months), at 12 months, 18 months and 24 months.

OUTCOME VARIABLES. Anthropometrical measures: Height, weight and waist-circumference, DXA-scans and bio-impedance measurements for determining the distribution of fat and muscle tissue. Physiological measures: Blood samples will be drawn in the morning after an overnight fast. Including measurements of total-cholesterol, HDL, LDL, TG, ASAT, ALAT, gamma-GT, bilirubin, creatinin, HbA1c and fasting insulin, c-peptide and glucose, TSH, fT4, CRP. Cortisol measurements from saliva and urine. Measurement of bloodpressure. Food records: The parents will be instructed to help their children to keep a diary of food and beverage intake for five days. They will use an electronic kitchen scale to weigh the food. Physical activity: Physical activity and sleep will be measured by using accelerometers. Psychological measures: The Child Behavior Checklist (CBCL) is a 138-item rating scale assessing behavioral and emotional symptoms in children/youth. Children's Depression Inventory (CDI). CDI is a 27-item self-report test assessing symptoms of depression in children (7-17 years). Self-Perception Profile for Children (SPPC). SPPC is a self-report measure of self-perception in children aged 8 to 14 years. The Dutch Eating Behavior Questionnaire Child version (DEBQ) is a measure of disturbed eating patterns in children and youth. The Youth Eating Disorder Examination-Questionnaire (YEDE-Q) is a self-reported measure of eating patterns and eating disorder psychopathology. OTHER MEASUREMENTS INCLUDED. The Parenting Scale (PS) is a 30-item questionnaire designed to measure different parental disciplines with children/youth. The scores on three sub-scales are calculated - Laxness, Overreactivity and Verbosity. The Barriers to Treatment Participation Scale (BTPS). The 44-item scale is developed and validated to address drop-out from treatment with out-patient psychological treatment of children and adolescents. Child and parent acceptability of the treatment will be measured by the FBSFT Acceptability Questionnaire.

STUDY AIMS:

1. To evaluate the effect of FBSFT compared to TAU for treatment of severe childhood and adolescent obesity in an ordinary health care setting on BMI, BMI SDS, body composition, cardio-metabolic health, eating habits, physical activity as well as psychological well-being.
2. To identify predictors of treatment success and treatment drop-out with a focus on family variables and mental health.
3. To evaluate treatment (FBSFT) implementation and treatment acceptability for children, parents and health care workers and experienced barriers to treatment, and how these factors influence children's and parents' treatment response.

ELIGIBILITY:
Inclusion Criteria:

* The sample will consist of children and adolescents (aged 6-18) referred to the Obesity Outpatient Clinic at Haukeland University Hospital by their general practitioner.
* Criteria for admission to the clinic is an (IOTF) isoBMI of > 35, or a isoBMI > 30 with obesity related co-morbidity.
* Both the child and at least one of the parents agrees to actively participate in the treatment.

Exclusion Criteria:

* Severe somatic or psychiatric illness that makes adherence to the treatment program impossible.
* Somatic conditions, syndromes or medications that lead to pathological weight gain.
* Participation in other obesity treatment programs.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in weight status, assessed as BMI, BMI standard deviation scores (SDSs) and percentages above the IOTF cut-off for overweight (%IOTF-25) | BMI will be measured at baseline and after 3, 6, 9, 12, 15, 18 and 24 months.
  Height, weight will be measured by trained assessors at the Obesity Outpatient Clinic.

SECONDARY OUTCOMES:
Change in waist circumference | Will be measured at baseline and after 3, 6, 9, 12, 15, 18 and 24 months.
  Will be measured by trained assessors at the Obesity Outpatient Clinic
Change in %body fat assessed by Bio-impedance | Measurements will be done at baseline, 6 months, 12 months, 18 months and 24 months
  Bio-impedance measurements of body composition will be conducted at the Obesity Outpatient Clinic using InBody 720.
Change in % body fat assessed by DXA | Measurements will be made at baseline, at 6 months, at 12 months, at 18 months and at 24 months.
  DXA-scans for determining the distribution of fat and muscle tissue will be conducted at the Department of Rheumathology at Haukeland University Hospital.
Change in Blood samples and cortisol measurements | measurements will be done at baseline, 6 months, 12 months, 18 months and 24 months
  Blood samples will be drawn in the morning after an overnight fast. Including measurements of total-cholesterol, HDL, LDL, TG, ASAT, ALAT, gamma-GT, bilirubin, creatinin, HbA1c and fasting insulin, c-peptide and glucose, TSH, fT4, CRP. Cortisol measurements from saliva and urine. A bio-bank for the storing and registering of biological materials is approved.
Change in blood pressure | Will be measured at baseline, 6 months, 12 months, 18 months and 24 months
  Blood pressure will be measured by the pediatrician at the obesity clinic
Changes in eating habits - Food diary | Measurements will be obtained at baseline, 6 months, 12, months, 18 months and 24 months
  The parents will be instructed to help their children to keep a diary of food and beverage intake for five days including two weekend days. They will use an electronic kitchen scale to weigh the food.
Changes in physical activity and sleep patterns - Accelerometers | Measurements will be made at baseline, 6 months, 12 months, 18 months and 24 months
  Physical activity and sleep patterns will be measured by using accelerometers. Accelerometers are small devices that register movement. The accelerometers that will be used in this study are worn on the non-dominant wrist and resemble a watch. The accelerometers record all uni-axial movement over 0.05G in one-minute epochs
Changes in psychological parameters - The Child Behavior Checklist (CBCL)/Youth self-report (YSR) | Measurements will be obtained at baseline, at 6 months, 12 months, 18 months and 24 months
  The Child Behavior Checklist (CBCL) is a 138-item rating scale assessing behavioural and emotional symptoms in children that has both a child/youth and parent form.
Changes in psychological parameters - Children's Depression Inventory (CDI) | Assessments at baseline, at 6 months, 12 months, 18 months and 24 months
  Children's Depression Inventory (CDI). CDI is a 27-item self-report test assessing the cognitive, affective and behavioural symptoms of depression in children (7-17 years).
Changes in psychological parameters - Self-Perception Profile for Children (SPPC). | Assessments at baseline, at 6 months, 12 months, 18 months and 24 months
  Self-Perception Profile for Children (SPPC). SPPC is a self-report measure of self-perception or self-esteem in children aged 8 to 14 years and is widely used for research purposes. The questionnaire includes 36 statements and the children are asked to evaluate to which degree the statement fits their thoughts about themselves.
Changes in eating habits - The Dutch Eating Behavior Questionnaire Child version (DEBQ) | Assessments at baseline, at 6 months, 12 months, 18 months and 24 months
  The Dutch Eating Behavior Questionnaire Child version (DEBQ) is a measure of disturbed eating patterns in children and youth (41). DEBQ consists of 3 sub-scales: emotional eating, external eating and restrained eating.
Changes in eating habits - The Youth Eating Disorder Examination-Questionnaire (YEDE-Q) | Assessments at baseline, at 6 months, 12 months, 18 months and 24 months
  The Youth Eating Disorder Examination-Questionnaire (YEDE-Q) is a self-reported measure of eating patterns and eating disorder psychopathology. The YEDE-Q was designed to include measurements of binge eating in youth which have been poorly covered in other self-report measures of eating pathology.

OTHER OUTCOMES:
The Parenting Scale (PS) | Assessment at baseline, 6 months, 12 months, 18 months and 24 months
  The Parenting Scale (PS) is a 30-item questionnaire designed to measure different parental disciplines with children and youth. The scores on three sub-scales are calculated - Laxness, Overreactivity and Verbosity.
The Barriers to Treatment Participation Scale (BTPS). | Assessment at 4 months after enrollment or point of deciding to end treatment for the FBSFT arm
  The Barriers to Treatment Participation Scale (BTPS). The 44-item scale is developed and validated to address drop-out from treatment with out-patient psychological treatment of children and adolescents. Scores are distributed across 4 sub-scales: (1) Stressors and obstacles that compete with treatment, (2) treatment demands and issues, (3) perceived relevance of the treatment, (4) therapeutic relationship.
FBSFT Acceptability Questionnaire. | Measurement at 6 months after enrollment for the FBSFT arm
  Child and parent acceptability of the treatment will be measured by the FBSFT Acceptability Questionnaire. The measure consists of two subscales: satisfaction and perceived utility. This measure has been informed by assessments used in a treatment study for pediatric obesity in the UK, which evaluates degree to which participants were pleased with the intervention and the extent to which they perceived components to be helpful

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Skjakodegard HF, Danielsen YS, Morken M, Linde SF, Kolko RP, Balantekin KN, Wilfley DE, Juliusson PB. Study Protocol: A randomized controlled trial evaluating the effect of family-based behavioral treatment of childhood and adolescent obesity-The FABO-study. BMC Public Health. 2016 Oct 21;16(1):1106. doi: 10.1186/s12889-016-3755-9. PMID 27769209